CLINICAL TRIAL: NCT00378105
Title: An Open-Label Phase I/II Study of the Safety and Efficacy of Bortezomib, Lenalidomide and Dexamethasone Combination Therapy for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Bortezomib, Lenalidomide and Dexamethasone Combination Therapy in Patients With Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Celgene Corporation (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Paul Richardson, MD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-150
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone

ARMS (1):
- lenalidomide, dexamethasone, bortezomib combination (Experimental): In this study each cycle will be 21 days and participants will begin the study medication in the clinic on Cycle 1 Day 1. Lenalidomide (capsules) will be taken daily for the first 2 weeks only (Day 1-14). Dexamethasone (tablets) will be taken on Day 1, 2, 4, 5, 8, 9, 11 and 12. Bortezomib will be given intravenously in the outpatient treatment clinic on Day 1, 4, 8 and 11. The third week is a rest period and no study medication will be given.
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Intravenously on days 1, 4, 8 and 11 of a 21 day cycle for a minimum of 8 cycles (dosage will vary depending upon when the participant enters the trial)
Drug: Lenalidomide — Taken orally twice a day for 2 weeks (days 1-14) of each 21-day cycle for a minimum of 8 cycles (dosage will vary depending upon when participant enters trial).
Drug: dexamethasone — Taken orally on days 1,2,4,5,8,9,11 of a 21-day cycle for a minimum of 8 cycles.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the bortezomib, lenalidomide and dexamethasone combination in patients with newly diagnosed multiple myeloma. We are looking for the highest dose of the combination that can be given safely and see how well it works as a combination in newly diagnosed patients.

DETAILED DESCRIPTION:
* The safe dose of dexamethasone is already known. The dose of bortezomib and lenalidomide will be increased during the study until the best and safest amount (or dose) is identified. The participant's dose of the study drugs will depend on when they enter the study.
* In this study each cycle will be 21 days and participants will begin the study medication in the clinic on Cycle 1 Day 1. Lenalidomide (capsules) will be taken daily for the first 2 weeks only (Day 1-14). Dexamethasone (tablets) will be taken on Day 1, 2, 4, 5, 8, 9, 11 and 12. Bortezomib will be given intravenously in the outpatient treatment clinic on Day 1, 4, 8 and 11. The third week is a rest period and no study medication will be given.
* During the course of the study treatment, tests and procedures will be performed at designated time periods. This includes; medical history updates, physical/neurological examinations, skeletal survey (x-rays or scan), blood samples, optional bone marrow aspiration/tissue biopsy, urine samples, 12-lead ECG, and MRI/CT scan (if needed).
* It is expected that study participants will receive study treatment for 8 cycles (168 days). If the participant completes the first 8 cycles of the study, has stable or responding disease and has not experienced bad side effects, they will be allowed to continue treatment on a maintenance schedule, detailed in the protocol, at the study doctor's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple myeloma based on standard diagnostic criteria or by the new International Myeloma Foundation 2003 Diagnostic Criteria
* Must not have been previously treated with any prior systemic therapy for the treatment of multiple myeloma
* Negative serum or urine pregnancy test
* Age 18 years or older
* Karnofsky performance status of greater or equal to 60

Exclusion Criteria:

* Greater or equal to Grade 2 peripheral neuropathy on clinical examination within 14 days before enrollment
* Renal insufficiency (serum creatinine >2.5 mg/dL)
* Evidence of mucosal or internal bleeding and/or platelet refractory
* ANC (absolute neutrophil count)< 1000 cells/mm3
* Hemoglobin < 8.0 g/dL
* AST (aspartate aminotransferase) or ALT (alanine aminotransferase) greater than or equal to 2 x ULN (upper limit of normal)
* Concomitant therapy medications that include corticosteroids
* Myocardial infarction within 6 months prior to enrollment according to NYHA (New York Heart Association) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Clinically relevant active infection or serious co-morbid medical conditions
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer
* Pregnant or breast-feeding
* Serious medical or psychiatric illness likely to interfere with participation in study
* Uncontrolled diabetes mellitus
* Hypersensitivity to acyclovir or similar anti-viral drug
* POEMS syndrome
* Known HIV infection
* Known active hepatitis B or C viral infection
* Known intolerance to steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Dytfeld D, Rosebeck S, Kandarpa M, Mayampurath A, Mellacheruvu D, Alonge MM, Ngoka L, Jasielec J, Richardson PG, Volchenboum S, Nesvizhskii AI, Sreekumar A, Jakubowiak AJ. Proteomic profiling of naive multiple myeloma patient plasma cells identifies pathways associated with favourable response to bortezomib-based treatment regimens. Br J Haematol. 2015 Jul;170(1):66-79. doi: 10.1111/bjh.13394. Epub 2015 Mar 30. PMID 25824111
- [Derived] Richardson PG, Weller E, Lonial S, Jakubowiak AJ, Jagannath S, Raje NS, Avigan DE, Xie W, Ghobrial IM, Schlossman RL, Mazumder A, Munshi NC, Vesole DH, Joyce R, Kaufman JL, Doss D, Warren DL, Lunde LE, Kaster S, Delaney C, Hideshima T, Mitsiades CS, Knight R, Esseltine DL, Anderson KC. Lenalidomide, bortezomib, and dexamethasone combination therapy in patients with newly diagnosed multiple myeloma. Blood. 2010 Aug 5;116(5):679-86. doi: 10.1182/blood-2010-02-268862. Epub 2010 Apr 12. PMID 20385792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 68 patients were enrolled in the United States. For the phase I part, this study enrolled 33 eligible patients between Sep13, 2006 and Aug16, 2007. For the phase II part, this study enrolled 35 eligible patients between Aug 20, 2007 and Feb18, 2008.
Pre-assignment Details: Participants were screened over a two-week period.
Groups:
- Phase 1 Population: Four levels of dose were evaluated and a standard 3+3 dose escalation schema was used to determine the MTD and additional patients were evaluated on the MTD level.
  1. Level 1 1 mg/m2/IV bortezomib daily Days 1,4, 8 and 11 40 mg PO dexamethasone daily Days 1, 2, 4, 5, 8, 9, 11, 12 and 15 mg/PO/day lenalidomide daily Days 1-14 followed by 7-day rest every 21 days
  2. Level 2 1.3 mg/m2/IV bortezomib daily Days 1,4, 8 and 11 40 mg PO dexamethasone daily Days 1, 2, 4, 5, 8, 9, 11, 12 and 15 mg/PO/day lenalidomide daily Days 1-14 followed by 7-day rest every 21 days
  3. Level 3 1.3 mg/m2/IV bortezomib daily Days 1,4, 8 and 11 40 mg PO dexamethasone daily Days 1, 2, 4, 5, 8, 9, 11, 12 and 20 mg/PO/day lenalidomide daily Days 1-14 followed by 7-day rest every 21 days
  4. Level 4 1.3 mg/m2/IV bortezomib daily Days 1,4, 8 and 11 40 mg PO dexamethasone daily Days 1, 2, 4, 5, 8, 9, 11, 12 and 25 mg/PO/day lenalidomide daily Days 1-14 followed by 7-day rest every 21 days
- Phase 2 Pupulation: Each subject received the maximum planned dose of 1.3 mg/m2/IV bortezomib daily Days 1, 4, 8 and 11 followed by a 10-day rest period, 20 mg PO dexamethasone single daily oral dose Days 1, 2, 4, 5, 8, 9, 11, 12 and25 mg/PO/QD (every day)lenalidomide daily Days 1-14 followed by 7-day rest every 21 days x 4 cycles and then at 10 mg/day on the same schedule for cycles 5 - 8. Each cycle of treatment consisted of 21 days.
Period: Overall Study
Arm/Group | Phase 1 Population | Phase 2 Pupulation
Started | 31 (Out of 33 enrolled, two patients went off study before start of therapy.) | 35
Completed | 11 | 5
Not Completed | 20 | 30
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Death | 1 | 0
Not completed — Going to transplant | 7 | 8
Not completed — Progressive disease | 3 | 3
Not completed — remain on study | 3 | 11
Not completed — Physician Decision | 0 | 2
Not completed — Going non-protocol therapy | 0 | 1
Not completed — necessity to increase lenalidomide dose | 0 | 1

BASELINE CHARACTERISTICS:
Population: The numbers excluded 2 patients who went off study prior to start of therapy (phase I part).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Population | Phase 2 Population | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Continuous [Median (Full Range); unit: years] | 57 [36 to 73] | 59 [22 to 86] | 58 [22 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate of the Drug Combination in This Patient Populations.
Description: Overall Response (OR) was defined as partial response (PR) or better. Response was assessed according to European Group for Blood and Marrow Transplant criteria, modified to include nCR and VGPR, from the International Uniform Response Criteria.
Time Frame: Full response assessment was conducted at the end of cycle 8 (average of168 days) and after cycle 4 (84 days) for patients proceeding to transplant.
Population: The numbers excluded 2 patients who went off study prior to start of therapy
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 Population | Phase II Population | Total
Number analyzed (Participants) | 31 | 35 | 66
percentage of participants | 100 [91 to 100] | 100 [92 to 100] | 100 [96 to 100]

2. Secondary Outcome: Estimated 18-month Progression Free Survival (PFS) Rate
Description: PD from European Bone Marrow Transplant (EBMT) Response Criteria Required one or more:
  >25% increased in the level of serum monoclonal paraprotein, which must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation, or >25% increased in 24-hour urinary light chain excretion (must also be an absolute increase of at least 200 mg/24 h and confirmed on a repeat investigation), or >25% increased in plasma cells in a bone marrow aspirate or biopsy (must also be an absolute increase of at least 10%) Definite increase in the size of existing lytic bone lesions or soft tissue plasmacytomas.
  Development of new bone lesions or soft tissue plasmacytomas (not including compression fracture).
  Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.8 mmol/L not attributable to any other cause).
  PFS was measured from treatment initiation to progression or death, censored at the date patients were last known to be alive and disease free
Time Frame: PFS rate at 18 months
Population: This numbers excluded 2 patients who went off study prior to start of therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 66
Percentage of participants | 75 [63 to 84]

3. Secondary Outcome: Percentage of Patients Who Remained in Response for More Than 18 Months
Description: Duration of response was measured from first response to progression or death, censored at the date patients were last known to be alive and disease free for patients who had not progressed or died.
Time Frame: Response rate at 18 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 66
Percentage of participants | 68 [55 to 79]

4. Secondary Outcome: Estimated 18-month Overall Survival Rate
Description: Overall survival was measured from treatment initiation to death, censored at the date patients were last known to be alive for those who had not died.
Time Frame: Survival rate at 18 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 66
Percentage of participants | 97 [88 to 99]

ADVERSE EVENTS:
Time Frame: Safety was assessed every cycle during the therapy.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 37/66
Other Adverse Events (participants affected / at risk) | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=66)
Sensory Neuropathy (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1
Rash/ desquamation (Skin and subcutaneous tissue disorders) | 1
Neuropathic pain (Nervous system disorders) | 2
Extremity Pain (General disorders) | 2
Insomnia (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Dizziness (General disorders) | 2
Motor Neuropathy (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 6
Anxiety (Psychiatric disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 9
Blurred Vision (Eye disorders) | 1
Elevated alanine transaminase (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Altered Mental Status (Psychiatric disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Pulmonary/ Upper Respiratory Event (Respiratory, thoracic and mediastinal disorders) | 2
Agitation (Psychiatric disorders) | 1
Altered Hearing (Ear and labyrinth disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Altered QTc interval (Cardiac disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 3
Elevated Creatinine (Metabolism and nutrition disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Infection (Infections and infestations) | 1
Stomach Hemorrhage (Vascular disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=66)
Sensory Neuropathy (Nervous system disorders) | 52
Fatigue (General disorders) | 40
Constipation (Gastrointestinal disorders) | 40
Peripheral Edema (Blood and lymphatic system disorders) | 30
Muscle Pain (Musculoskeletal and connective tissue disorders) | 28
Rash/desquamation (Skin and subcutaneous tissue disorders) | 23
Diarrhea (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 21
Neuropathic Pain (Nervous system disorders) | 19
Extremity pain (Nervous system disorders) | 18
Insomnia (General disorders) | 19
Hyperglycemia (Metabolism and nutrition disorders) | 17
Dizziness (General disorders) | 15
Other Constitutional Event (General disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Motor Neuropathy (Nervous system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Pruritis/itching (Skin and subcutaneous tissue disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 4
Anxiety (Psychiatric disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Blurred Vision (Eye disorders) | 8
Elevated Alanine Transaminase (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 4
Altered mental status (Psychiatric disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Pulmonary/upper respiratory event (Respiratory, thoracic and mediastinal disorders) | 4
Agitation (Psychiatric disorders) | 3
Altered hearing (Ear and labyrinth disorders) | 3
Anemia (Blood and lymphatic system disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9
bloating (Gastrointestinal disorders) | 9
joint pain (Musculoskeletal and connective tissue disorders) | 9
anorexia (Metabolism and nutrition disorders) | 8
dysgeusia (Nervous system disorders) | 8
tremor (Nervous system disorders) | 8
cognitive disturbance (Nervous system disorders) | 8
infection (Infections and infestations) | 10
metabolic lab disorder (Metabolism and nutrition disorders) | 13
tinnitus (Ear and labyrinth disorders) | 7
dysarthria (Nervous system disorders) | 7
bone pain (Musculoskeletal and connective tissue disorders) | 6
cough (Respiratory, thoracic and mediastinal disorders) | 6
cushingoid appearance (Endocrine disorders) | 6
depression (Nervous system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 6
headache (Nervous system disorders) | 6
hypocalcemia (Metabolism and nutrition disorders) | 6
sweating (Skin and subcutaneous tissue disorders) | 6
head and neck edema (General disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Alkaline phosphatase increased (Investigations) | 4
dry eye (Eye disorders) | 4
Genital and trunk edema (General disorders) | 4
flushing (Vascular disorders) | 4
hypomagnesemia (Metabolism and nutrition disorders) | 4
hypotension (Vascular disorders) | 4
personality change (Psychiatric disorders) | 4
chills (General disorders) | 4
vomiting (Gastrointestinal disorders) | 4
weight gain (Investigations) | 4
confusion (Psychiatric disorders) | 3
gait disturbance (General disorders) | 3
gastritis (Gastrointestinal disorders) | 3
neck pain (Musculoskeletal and connective tissue disorders) | 3
urinary frequency (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days